CLINICAL TRIAL: NCT03995628
Title: Randomized, Controlled Trial of Post-operative Steroids and Pain Control After Tonsillectomy
Brief Title: Steroids and Pain Control After Tonsillectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Phayvanh Pecha, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00081346
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-07

CONDITIONS: Tonsillitis; Obstructive Sleep Apnea of Child
MeSH Terms: conditions — Tonsillitis | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Steroid Group (Experimental): Participants will receive a one-time dose of oral dexamethasone at 0.5 mg/kg on the third post-operative day
  Interventions: Drug: Dexamethasone
- No Steroid Group (Placebo Comparator): Participants will receive placebo on third post-operative day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — One dose of dexamethasone (0.5 mg/kg) on post-operative day 3 after tonsillectomy
  Other Names: Decadron
  Arms: Steroid Group
Drug: Placebo — One dose of placebo on post-operative day 3 after tonsillectomy
  Arms: No Steroid Group

SUMMARY:
This research study aims to find out if a single oral dose of steroid after tonsillectomy will reduce pain and decrease the need for narcotic medications.

DETAILED DESCRIPTION:
The study will be performed prospectively and in a randomized, double-blinded, placebo controlled manner. Patients meeting inclusion and not violating exclusion criteria will be randomized to either receive a single oral steroid dose or a single placebo dose on the third day after surgery. All study patients will otherwise receive the standard of care in all other aspects of their treatment. That is, the surgery itself, the post-operative pain control strategies/medication, patient instructions, and follow up will not differ between the two groups. The pediatric otolaryngology department has standardized post-operative pain control (a specific order set is used) which will ensure no differences between different providers.

Oral dexamethasone is the study drug and will be given in 0.5mg/kg dosage and the route is 3mg capsules in increments of one capsule. Doses are calculated by weight and rounded up to the nearest 3mg up to a maximum of 12mg (4 capsules). Parents are instructed to give the medication on the morning of the third day after surgery. Parents can either have the child swallow the capsule or, if the child does not tolerate this, open the capsule and mix the contents into food the consistency of applesauce, then administer. A placebo will also be designed in the same route as the oral dexamethasone. Both the placebo and oral dexamethasone capsules will be purchased from by Tidewater Pharmacy and Compounding, an accredited pharmacy located in Mt. Pleasant, South Carolina12. Weight based instructions will be included with the study materials. During distribution, the member of the study team delivering the study materials will confirm the dosing with the parents.

Study materials will be assembled and randomized by the project lead, and will include a small container with four capsules of either placebo or oral dexamethasone. All study materials will be assigned a unique record number between 001 and 150. The materials will be block-randomized in groups of 30 to either contain placebo or oral dexamethasone, and linked to the record number in a secured file held by the project lead. This file will be inaccessible to any but the project lead during data collection. The study materials with the drug or placebo will be kept in a temperature controlled locked cabinet at the study site, MUSC Children's Health R. Keith Summey Medical Pavilion.

Immediately following the procedure in the operating room, once lack of exclusion criteria has been confirmed by the operating surgeon, patients will be assigned a subject record number in numerical order. This record number will be recorded, linked to the patient's medical record number, and kept in a secure file separate from the randomization list. The randomization process will be blinded from the parents, subjects, study coordinator, and operating surgeon. The subject's parents will then receive study materials that correspond to their unique record number, which will include either four 3mg dexamethasone capsules or four placebo capsules. Weight based instructions will be included with this dosing, and providers and/or research team members will go over these instructions with parents again when giving the study materials.

After randomization, the operating surgeon will complete a questionnaire to document details of the surgery, including: who performed the surgery, intracapsular versus extracapsular tonsillectomy, estimated blood loss, and use of suction cautery on the tonsillar bed. This will be collected by the study coordinator and linked to the patient record number.

Patients enrolled in the study will receive a "post-operative pain and medication diary" upon discharge from their procedure. Patients (parents) will be instructed to record daily pain control (on a validated visual analog scale (VAS)) and daily medication administration (opioid and non-opioid analgesic) for post-operative days 0-6 in this diary. Patients will return the diary to the study team via email, fax, text message, or a pre-addressed, stamped envelope. Reminders to return the materials will be sent to the parents periodically by the study coordinator via email, text message, or phone call. Recall bias will be reduced by the incorporation of the diary to aid parents' memory. The study coordinator will transcribe pain control and medication consumption data into the REDCap data compilation system.

The Faces Pain Scale-Revised13 will be used to assess patient pain on post-operative day 0-6. The scale will be provided to the patient in their discharge packet and a diary to record daily pain score will be provided. Mean VAS for post-operative day 1-3 and mean VAS for post-operative day 4-6 will be calculated for comparison.

Daily medication administration will be recorded by parents, specifically the number of doses of opioid and non-opioid analgesic medication consumed. For opioids, doses consumed will be cross-referenced against the weight-based dose prescribed in order to calculate daily oral morphine equivalents (OME) consumed. Mean daily OME will be calculated for post-operative day 1-3 and for post-operative day 4-6 for comparison.

At 30-days following surgery, participant patient charts will be queried by the study coordinator for presentation to the emergency room, readmission, and oropharyngeal hemorrhage. Presentation to the emergency room and readmission will be included if considered related to the procedure. Related emergency room presentation or readmission is defined as that due to throat pain, neck pain, ear pain, poor oral intake due to pain, dehydration due to poor oral intake caused by pain, and bleeding from the mouth or nose. Regarding oropharyngeal hemorrhage, any subjective or objective bleeding from the mouth or nose within 30 days of the procedure will be considered related to the procedure. Oropharyngeal hemorrhage will be divided into three groups: mild (not requiring admission, manifested as phone call or presentation to the emergency room), moderate (requiring admission but not return to the operating room), and severe (requiring urgent or emergent intubation and/or control of hemorrhage in the operating room).

If patients are experiencing pain uncontrolled by oral medications after tonsillectomy, providers at our institution will occasionally choose to give a dose of steroids prior to the third postoperative day or a second dose of steroids after the third postoperative day to help with pain control. If study patients have pain prior to the third postoperative day and a provider believes steroids are indicated, the patient should be given this medication, and then will be instructed not to take the study medication and will be excluded from analysis. If patients have pain on the third postoperative day and have already taken the study medication, they will be instructed to wait at least 6 hours before receiving another dose of steroids. All of this will be discussed in detail when obtaining consent, and will be included in the study materials given to parents.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-12
* Tonsillectomy with or without adenoidectomy for any indication
* Outpatient (same day) surgery

Exclusion Criteria:

* Bleeding disorder
* Intra-operative surgical or anesthetic complication or unplanned admission
* Pre-operative steroid use (defined as any steroid use greater than three days duration within 30 days prior to tonsillectomy)
* Pre-operative opioid use (defined as any opioid use within 30 days prior to tonsillectomy)
* Inability of parent/guardian to be contacted by phone for follow up
* Inability or unwillingness of subject or legal guardian/representative to give informed consent

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 163 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Mean Visual Analog Score of Pain | Postoperative day 6
  On postoperative days 0-6, the caregiver assesses participant pain using The Faces Pain Scale-Revised, which measures pain via a visual analog score. The visual analog score is an integer value between 0-10, where 0 represents no pain and 10 represents maximum pain. The mean visual analog score on postoperative day 1-3 and the mean visual analog score on postoperative day 4-6 will be calculated for comparison between arms of the study. Lower mean visual analog scores on days 4-6 represent a better outcome.

SECONDARY OUTCOMES:
Mean Opioid Consumption | Postoperative day 6
  The caregiver will keep a log of daily doses of opioids given to the participant for postoperative days 0-6. The mean total opioid consumption on postoperative day 1-3 and mean total opioid consumption on postoperative day 4-6 will be calculated for comparison between arms of the study.
Mean NSAID and Acetaminophen Consumption | Postoperative day 6
  The caregiver will keep a log of daily doses of NSAIDs and/or acetaminophen given to the participant for postoperative days 0-6. The mean total NSAID and acetaminophen consumption on postoperative day 1-3 and on postoperative day 4-6 will be calculated for comparison between arms of the study.
Rate of Nausea and Vomiting | Postoperative day 6
  The caregiver will keep a daily log of of the participant's nausea and vomiting status for postoperative days 0-6. The mean total instances of nausea and vomiting on postoperative day 1-3 and on postoperative day 4-6 will be calculated for comparison between arms of the study.
Diet and Activity Levels | Postoperative day 6
  The caregiver will keep a daily log of of the participant's diet and activity levels for postoperative days 0-6. The mean diet and activity levels on postoperative day 1-3 and on postoperative day 4-6 will be calculated for comparison between arms of the study.
Rate of 30-Day Readmission | Postoperative day 30
  A chart review will be performed to assess whether the participant ever needed to be readmitted to the hospital for postoperative complications, pain control, or dehydration due to poor oral intake within the first 30 days after surgery.
Rate of 30-Day Emergency Room Visits | Postoperative day 30
  A chart review will be performed to assess whether the participant ever presented to the emergency room for postoperative complications, pain control, or dehydration due to poor oral intake within the first 30 days after surgery.
Rate of Postoperative Oropharyngeal Hemorrhage | Postoperative day 30
  A chart review will be performed to assess whether postoperative oropharyngeal hemorrhage occurred in the 30 days following surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Phayvanh Pecha, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

REFERENCES:
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329
- [Background] Tan GX, Tunkel DE. Control of Pain After Tonsillectomy in Children: A Review. JAMA Otolaryngol Head Neck Surg. 2017 Sep 1;143(9):937-942. doi: 10.1001/jamaoto.2017.0845. PMID 28662233
- [Background] Batistaki C, Kaminiotis E, Papadimos T, Kostopanagiotou G. A Narrative Review of the Evidence on the Efficacy of Dexamethasone on Postoperative Analgesic Consumption. Clin J Pain. 2017 Nov;33(11):1037-1046. doi: 10.1097/AJP.0000000000000486. PMID 28177939
- [Background] Vlok R, Melhuish TM, Chong C, Ryan T, White LD. Adjuncts to local anaesthetics in tonsillectomy: a systematic review and meta-analysis. J Anesth. 2017 Aug;31(4):608-616. doi: 10.1007/s00540-017-2310-x. Epub 2017 Jan 24. PMID 28120104
- [Background] Redmann AJ, Maksimoski M, Brumbaugh C, Ishman SL. The effect of postoperative steroids on post-tonsillectomy pain and need for postoperative physician contact. Laryngoscope. 2018 Sep;128(9):2187-2192. doi: 10.1002/lary.27167. Epub 2018 Mar 24. PMID 29573428
- [Background] Rosen HI, Bergh IH, Oden A, Martensson LB. Patients experiences of pain following day surgery - at 48 hours, seven days and three months. Open Nurs J. 2011;5:52-9. doi: 10.2174/1874434601105010052. Epub 2011 Jul 6. PMID 21769308
- [Background] Cronin J, Kennedy U, McCoy S, An Fhaili SN, Crispino-O'Connell G, Hayden J, Wakai A, Walsh S, O'Sullivan R. Single dose oral dexamethasone versus multi-dose prednisolone in the treatment of acute exacerbations of asthma in children who attend the emergency department: study protocol for a randomized controlled trial. Trials. 2012 Aug 21;13:141. doi: 10.1186/1745-6215-13-141. PMID 22909281